CLINICAL TRIAL: NCT01494935
Title: Effect of High Fat and High Glycemic Diets on Muscle Protein Synthesis in Somali Immigrants and Americans of Northern European Descent
Brief Title: "Effect of High Fat and High Glycemic Diets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, K. Sreekumaran Nair, MD, Mayo Clinic
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 10-005948
Record Dates: First submitted 2011-11-18; First posted 2011-12-19 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (2):
- Normal glycemic diet (Experimental): COntrol diet with fat and glycemic index similar to typical American diet.
  Interventions: Behavioral: Control diet
- High-fat, high-glycemic diet (Experimental): High-fat, high-glycemic diet
  Interventions: Behavioral: High Glycemic Diet

INTERVENTIONS:
Behavioral: High Glycemic Diet — NORMAL FAT AND GLYCEMIC DIET CONSUMED High FAT AND Glycemic Diet consumed
  Arms: High-fat, high-glycemic diet
Behavioral: Control diet — Normal fat, normal fat diet
  Arms: Normal glycemic diet

SUMMARY:
The investigators will determine whether people with high muscle mitochondrial capacity produce higher amount of reactive oxygen species (ROS) on consuming high fat /high glycemic diet and thus exhibit elevated cellular oxidative damage. The investigators previously found that Asian Indian immigrants have high mitochondrial capacity in spite of severe insulin resistance. Somalians are another new immigrant population with rapidly increasing prevalence of diabetes. Both of these groups traditionally consume low caloric density diets, and the investigators hypothesize that when these groups are exposed to high-calorie Western diets, they exhibit increased oxidative stress, oxidative damage, and insulin resistance. The investigators will compare Somalians and NE Americans who are matched for age, BMI, and sex. The investigators will measure ROS production in skeletal muscle following high fat/high glycemic diet vs. healthy diet. The investigators will compare the oxidative damage to proteins, DNA, and lipids in these two populations following 10 days of high fat/high glycemic index diet in comparison with low fat diet. The investigators will determine if elevated levels of oxidative damage in Somali immigrant populations is accompanied by high mitochondrial capacity, higher ROS-emitting potential, and lower insulin sensitivity than NE. The proposed study will be performed utilizing the state-of-the-art proteomic and metabolomic methods many of which were recently developed in our laboratory. The investigators expect the results from this study to provide seminal insights into the underlying mechanism of insulin resistance and type 2 diabetes, in addition to demonstrating mechanisms by which a functional proteome is maintained in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Somali immigrants age 40-65,
* BMI 23-34 kg/m2,
* sedentary (exercise less than 2 days per week for less than 20 minutes).

Inclusion criteria:

* for Northern European descendants same as for Somali immigrants plus need to match a Somali immigrant for age, BMI and habitual activity.

Exclusion Criteria:

* Triglycerides on screening examination of greater than 300;
* pregnant or lactating women.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-04; Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | Measured at day 0 (baseline) and day 10 (of high fat meals)
  The investigators will determine the change from baseline in insulin sensitivity using a hyperinsulinemic euglycemic clamp. Measurments will be performed at baseline and following 10 days of exercise a high fat diet.

SECONDARY OUTCOMES:
ceramides and diacylglycerol | Measured at day 0 (baseline) and day 10 (of high fat meals)
  The investigators will determine the change from baseline in skeletal insulin ceramide and diacylglycerol concentrations. Measurments will be performed at baseline and following 10 days of exercise a high fat diet.

CONTACTS AND LOCATIONS:
Overall Officials: Sreekumaran Nair, MD, Ph.D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials